CLINICAL TRIAL: NCT02739139
Title: Randomized Double-blind, Placebo-Controlled, Parallel Group, Efficacy Study of AlphaBRAIN(TM) Administered Orally
Brief Title: Efficacy Study of AlphaBRAIN Administered Orally
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Onnits Labs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB-001
Record Dates: First submitted 2013-09-25; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Cognitive Functioning

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: AlphaBrain
- AlphaBrain (Experimental): AlphaBrain(TM)
  Interventions: Dietary Supplement: AlphaBrain

INTERVENTIONS:
Dietary Supplement: AlphaBrain — Alpha BRAIN® (Onnit Labs LLC) is a multi-ingredient nutritional supplement that purports to enhance cognitive function in healthy adults. The commercially available product contains 12 naturally occurring compounds

SUMMARY:
The manufacturers of AlphaBRAIN(TM) claim that their product, when taken as directed, has beneficial effects on cognition. The active ingredient in AlphaBRAIN, Huperzine A, is a naturally occurring compound found in firmoss and also thought to be an acetylcholinesterase inhibitor. Numerous clinical studies have been undertaken to investigate the effects of Huperzine A on cognition and have demonstrated benefit to cognition in both individuals diagnosed with neurodegenerative diseases as well as performance on academic tasks by students. However, to our knowledge, there are no randomized controlled trials evaluating the effects of AlphaBRAIN(TM) on cognition. Thus, the purpose of the current study is to assess the effects of daily oral administration of AlphaBRAIN(TM) on cognitive functioning, as compared to placebo, after 45 days of treatment.

1. To evaluate a single daily dose of AlphaBRAIN(TM) vs placebo given orally on the change in a battery of standardized neuropsychological tests (see attached).
2. A secondary objective is to evaluate a single daily dose of AlphaBRAIN(TM) vs placebo given orally on sleep.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling and can provide informed consent.
* MMSE score of ≥ 26.
* Body Mass Index within two standard deviations of the norm.
* Fluent in English.
* Willing to complete all study assessments.
* Adequate visual and auditory acuity to allow for neuropsychological testing.

Exclusion Criteria:

* MMSE score < 26
* Body Mass Index greater then two standard deviations from the norm.
* Visual or Auditory disability which would interfere with neuropsychological testing.
* No past diagnosis of Stroke, ADD/ADHD, Learning Disability or Cardiac Condition.
* No current life threatening illnesses.
* Not currently (past 60 days) taking antidepressants or other psychoactive medications.
* Not currently taking any non-prescription cognitive enhancers (nutraceuticals or vitamins such as Ginko biloba.
* No history of alcohol or drug or dependence as defined by the DSM-IV-TR.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Performance on Standardized Neuropsychological Battery (Verbal Memory; Executive Functioning; Visual Memory; Working Memory; Attention; Processing Speed) | Six Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Center for Memory, Chestnut Hill, Massachusetts, United States